CLINICAL TRIAL: NCT02894697
Title: Clinical Significance of Pre-interventional Optical Coherence Tomography in Bioresorbable Vascular Scaffold Implantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a problem with the supply and demand of the stent used in the study, it is difficult to register the target so the study ends early.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2016-0038
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Angiography-guidance (Active Comparator)
  Interventions: Device: Angiography-guided PCI with BVS
- OCT-guidance (Experimental)
  Interventions: Device: Optical coherence tomography-guided PCI with BVS

INTERVENTIONS:
Device: Angiography-guided PCI with BVS — Everolimus-eluting bioresorbable vascular scaffold (Absorb, Abbott Vascular, Santa Clara, CA, USA) was made from a bioabsorbable polylactic acid backbone which is coated with a more rapidly absorbed polylactic acid layer that contains and controls the release of the antiproliferative drug, everolimus. PCI will be performed with BVS under conventional coronary angiography without any other intravascular imaging modality. After PCI, postprocedural OCT will be evaluated to find OCT-defined suboptimal results requiring additional PCI. If there is OCT-defined suboptimization, additional PCI will be performed including balloon angioplasty or additional stent or BVS implantation for scaffold optimization. Further postprocedural OCT will be also evaluated whether scaffold implantation is fully optimized or not.
  Arms: Angiography-guidance
Device: Optical coherence tomography-guided PCI with BVS — Everolimus-eluting bioresorbable vascular scaffold (Absorb, Abbott Vascular, Santa Clara, CA, USA) was made from a bioabsorbable polylactic acid backbone which is coated with a more rapidly absorbed polylactic acid layer that contains and controls the release of the antiproliferative drug, everolimus. For optimized PCI, both conventional coronary angiography and optical coherence tomography can be used before stent implantation. After PCI, postprocedural OCT will be evaluated to find OCT-defined suboptimal results requiring additional PCI. If there is OCT-defined suboptimization, additional PCI will be performed including balloon angioplasty or additional stent or BVS implantation for scaffold optimization. Further postprocedural OCT will be also evaluated whether scaffold implantation is fully optimized or not.
  Arms: OCT-guidance

SUMMARY:
Previous studies reported 20-30% of under-expansion or malapposition with BVS, which would increase the risk of adverse events including late stent thrombosis. OCT-guidance may improve more optimized scaffold placement and also better outcomes. However, there is still no sufficient evidence that OCT has an inevitable role in optimal implantation of BVS and it should be more evaluated in real practice. In the study, the investigators will evaluate an incidence of OCT-defined BVS sub-optimization requiring additional PCI+A1.

DETAILED DESCRIPTION:
It is well-known that non-optimal stent implantation associated with under-expansion or incomplete strut apposition during percutaneous coronary intervention (PCI) leads to a higher incidence of restenosis and stent thrombosis. OCT-guided PCI with metallic stent has previously been shown to be safe and feasible, resulting in better clinical outcomes compared with angiography-only guided PCI. Everolimus-eluting bioabsorbable vascular scaffold (BVS; Abbott Vascular, Santa Clara, CA, USA) was made from a bioabsorbable polylactic acid backbone which is coated with a more rapidly absorbed polylactic acid layer that contains and controls the release of the antiproliferative drug, everolimus. BVS has a number of proposed advantages over current metallic stent technology. These include elimination of chronic sources of vessel irritation and inflammation, which can reduce the potential risk of late scaffold thrombosis after complete scaffold bioresorption. Although the current generation of the Absorb BVS have larger strut thickness of 150 μm compared with 80 μm of strut of Xience stent, the acute recoil of the polymeric device was similar to that of metallic stent. However, operators tented to use dilating devices less aggressively because of the concerns about limitation in elongation-at-break of polylactide.

Previous studies reported 20-30% of under-expansion or malapposition with BVS, which would increase the risk of adverse events including late stent thrombosis. OCT-guidance may improve more optimized scaffold placement and also better outcomes. However, there is still no sufficient evidence that OCT has an inevitable role in optimal implantation of BVS and it should be more evaluated in real practice. In the study, the investigators will evaluate an incidence of OCT-defined BVS sub-optimization requiring additional PCI+A1.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Patients with ischemic heart disease who are considered for coronary revascularization with PCI
* Significant coronary de novo lesion (stenosis > 70% by quantitative angiographic analysis) treated by single BVS ≤ 28 mm
* Reference vessel diameter of 2.5 to 3.5 mm by operator assessment

Exclusion Criteria:

* Complex lesion morphologies such as aorto-ostial, unprotected left main, chronic total occlusion, graft, thrombosis, and restenosis
* Contraindication or hypersensitivity to anti-platelet agents or contrast media
* Creatinine level ≥ 2.0 mg/dL or ESRD
* Severe hepatic dysfunction (3 times normal reference values)
* Pregnant women or women with potential childbearing
* Inability to understand or read the informed content

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
An incidence of OCT-defined suboptimization of BVS requiring additional BVS | 1 second after angiographic scaffold optimization is obtained
  An incidence of OCT-defined BVS suboptimization requiring additional PCI
  : A composite of minimal scaffold area <5 mm2, residual area stenosis >20%, major edge dissections, incomplete strut apposition and scaffold pattern disruptions

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SY, Kang DY, Hong SJ, Ahn JM, Ahn CM, Park DW, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Park SJ, Hong MK. Optical Coherence Tomography for Coronary Bioresorbable Vascular Scaffold Implantation: A Randomized Controlled Trial. Circ Cardiovasc Interv. 2020 Jan;13(1):e008383. doi: 10.1161/CIRCINTERVENTIONS.119.008383. Epub 2020 Jan 9. PMID 32525410